CLINICAL TRIAL: NCT01796704
Title: Comparison of the Prediction Derived by the Cardiovascular Performance Reserve Index (Calculated From Physiological Parameters) With the Clinical Evaluation
Brief Title: Comparison of the Prediction Derived by the Cardiovascular Performance Reserve Index With the Clinical Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: COM120018CTIL
Record Dates: First submitted 2013-01-29; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2012-10

CONDITIONS: Healthy; Heart Failure
Keywords: functional capacity; NYHA class
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy and mild heart failure: diversity of patients

SUMMARY:
The study hypothesizes that an assumed cardiovascular performance reserve is physiologically detectable.

High reserve at rest characterizes a healthy person while low reserve at rest characterizes low functional capacity e.g. heart failure. The lower the reserve the severer the morbidity.

The reserve may be estimated through CVRI (cardiovascular reserve index) which is computed by an algorithm composed of physiological measurements taken during the patient visit.

In this study the investigators evaluate CVRI capability in prediction of functional capacity in comparison with the clinical evaluation during the same visit.

DETAILED DESCRIPTION:
The study hypothesizes that an assumed cardiovascular performance reserve is physiologically detectable and continuously monitored by a physiological control (reserve control)not yet discovered.

High reserve at rest characterizes a healthy person while low reserve at rest characterizes low functional capacity e.g. heart failure. The lower the reserve the severer the morbidity.

The reserve is decreased reversibly with aerobic activity and may reach an exhaustion threshold in which the assumed reserve control induces a reversible fatigue and dyspnea which dissolve once the activity decreased.

The reserve may be estimated through CVRI (cardiovascular reserve index) which is computed by an algorithm composed of physiological measurements taken during the patient visit (composed of blood pressure, heart rate, respiratory rate, central venous pressure or its estimation, weight, height and gender.

In this study the investigators evaluate CVRI capability in prediction of functional capacity in comparison with the clinical evaluation during the same visit (cross sectional comparison).

ELIGIBILITY:
Inclusion Criteria:

* adult informed consent

Exclusion Criteria:

* an emergency case

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adults both genders:
  healthy subjects visiting for administrative cause healthy subject during acute illness patients with chronic conditions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
cardiovascular reserve index | 1 day
  CVRI

CONTACTS AND LOCATIONS:
Overall Officials: Uri Gabbay, M.D, M.P.H., Principal Investigator — Tel Aviv University
Locations (1):
- Independent physician Clinic Clalit Health Services, Tel Aviv, Israel